CLINICAL TRIAL: NCT03720392
Title: A Phase 2 Study of Fecal Microbiota Transplantation (FMT) in Recipients After Allogeneic Hematopoietic Cell Transplantation (HCT)
Brief Title: Fecal Microbiota Transplantation (FMT) in Recipients After Allogeneic Hematopoietic Cell Transplantation (HCT)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to sponsor decision
Sponsor: Zachariah Michael DeFilipp (Other)
Responsible Party: Sponsor-Investigator, Zachariah Michael DeFilipp, Principal Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-293
Record Dates: First submitted 2018-10-24; First posted 2018-10-25 (Actual); Results first posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Allogeneic Hematopoietic Cell Transplantation (HCT)
Keywords: Allogeneic Hematopoietic Cell Transplantation (HCT)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FMT Capsules (Experimental): * Two doses of FMT: one standard dose starting within four (4) days from the start of the conditioning regimen prior to HCT and one non-standard dose starting within 4 weeks after engraftment after HCT.
  * A standard dose of oral FMT is 15 capsules per day for two consecutive days,
  Interventions: Drug: FMT
- Placebo Capsules (Placebo Comparator): * Two doses of placebo, instead of FMT: one starting within four (4) days from the start of the conditioning regimen prior to HCT and the second one starting within 4 weeks after engraftment after HCT.
  * A standard dose of oral Placebo is 15 capsules per day for two consecutive days,
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FMT — FMT is a process utilizing microbial components which are the good, healthy bacteria that would otherwise naturally occur in the body.
  Arms: FMT Capsules
Drug: Placebo — a harmless pill, medicine, or procedure prescribed more for the psychological benefit to the patient than for any physiological effect.
  Arms: Placebo Capsules

SUMMARY:
This research study is studying the role fecal microbiota transplantation may play in post-Hematopoietic Cell Transplantation (HCT) recipients

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved FMT for this use.

After HCT, the body's microbiome (the natural existence of various bacteria and organisms) in the intestinal tract may be affected, in that the number and types of good bacteria is reduced (also called a reduction in microbial flora diversity). Studies have shown that the number and types of good bacteria in the gut can impact whether or not a person develop a disease called graft-versus-host disease (GVHD). GVHD occurs when donated bone marrow cells attack the body with an immune response. Researchers believe that more microbial flora diversity in the gut is linked to a lower risk of developing GVHD.

FMT is a process utilizing microbial components which are the good, healthy bacteria that would otherwise naturally occur in the body. Since the participant may have decreased microbial flora diversity after HCT, these microbial components are taken from a 3rd party donor. They are extracted from fecal matter (stool) and put into a capsule which the participant then ingest.

Researchers believe that FMT administration may play a role in restoring higher microbial flora diversity in the gut. Therefore, FMT administration may play a role in decreasing the likelihood of developing GVHD.

In this research study, the investigators are...

* Examining the microbial flora diversity of your gut after FMT administration
* Looking for incidence rate of GVHD and other post-HCT complications

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 18 and ≤ 80 years old
* Patients designated to undergo myeloablative or intermediate intensity allogeneic peripheral blood or bone marrow hematopoietic cell transplantation. Consent will be obtained prior to admission for HSCT. Patients receiving any donor source of stem cells are eligible. Eligible conditioning regimens are those defined as myeloablative by the ASBMT Consensus Criteria (Bacigalupo 2009) as well as the combination of fludarabine with melphalan (100-140 mg/mg2)
* Any GVHD prophylaxis regimen is allowed.
* ECOG performance status ≤ 2 (Karnofsky ≥ 60%, see Appendix A)
* Patients with adequate physical function as measured by

  * Cardiac: Left ventricular ejection fraction at rest must be ≥ 40%, or shortening fraction >25%
  * Hepatic:
  * Bilirubin ≤ 2.5 mg/dL, except for patients with Gilbert's syndrome or hemolysis
  * ALT, AST, and Alkaline Phosphatase < 5 x ULN
  * Renal: Serum creatinine within normal range, or if serum creatinine is outside normal range, then renal function (measured or estimated creatinine clearance or GFR) ≥ 40mL/min/1.73m2
  * Pulmonary: DLCO (corrected for hemoglobin), FEV1 and FVC ≥ 50% predicted
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Women of childbearing potential will have a urine pregnancy test, which must be negative, on Study Day 1, prior to receiving FMT. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study and for 3 months after FMT.
* Ability to understand and the willingness to sign a written informed consent document, including the willingness to accept risk of unrelated donor stool.
* Ability to swallow large capsules.

Exclusion Criteria:

* Prior allogeneic hematopoietic stem cell transplantation. (Patients may have received a prior autologous hematopoietic stem cell transplant.)
* Participants who are receiving any other investigational agents.
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with active or uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
* Planned use of prophylactic donor lymphocyte infusion (DLI) therapy.
* Delayed gastric emptying syndrome or large hiatal hernia
* Known chronic aspiration
* Participants with a history of significant allergy to foods not excluded from the donor diet (excluded foods are tree nuts, peanuts, shellfish, eggs)
* Pregnant and breast-feeding women are ineligible because they are not eligible for hematopoietic stem cell transplantation.
* HIV-positive participants are ineligible.
* Participants who are unable to swallow pills.
* Participants with end-stage liver disease (cirrhosis)
* Participants with acute, active gastrointestinal infection (e.g., typhlitis, diverticulitis, appendicitis)
* Participants with inflammatory bowel disease (e.g., ulcerative colitis, Crohn's)
* Prior total colectomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zachariah DeFilipp, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 2 participants who withdrew from the trial prior to randomization thus not evaluable.
Groups:
- FMT Capsules: * Two doses of FMT: one standard dose starting within four (4) days from the start of the conditioning regimen prior to HCT and one non-standard dose starting within 4 weeks after engraftment after HCT.
  * A standard dose of oral FMT is 15 capsules per day for two consecutive days,
  FMT: FMT is a process utilizing microbial components which are the good, healthy bacteria that would otherwise naturally occur in the body.
- Placebo Capsules: * Two doses of placebo, instead of FMT: one starting within four (4) days from the start of the conditioning regimen prior to HCT and the second one starting within 4 weeks after engraftment after HCT.
  * A standard dose of oral Placebo is 15 capsules per day for two consecutive days,
  Placebo: a harmless pill, medicine, or procedure prescribed more for the psychological benefit to the patient than for any physiological effect.
Period: Overall Study
Arm/Group | FMT Capsules | Placebo Capsules
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FMT Capsules | Placebo Capsules | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients Who Achieve Gut Microbiome Diversity at One Month Following the Final Post-HCT FMT
Description: Gut microbiome diversity will be assessed using urinary 3-indoxyl sulfate (3-IS) levels, with 35 umol/mmol creatinine as the cutoff (≥ 35: diverse; < 35: not diverse).
Time Frame: 1 Month
Population: No analyses for this primary outcome were performed because the study was terminated after only 6 treated patients and there were only a few samples collected.
Arm/Group | FMT Capsules | Placebo Capsules
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants With Acute Graft-Versus-Host-Disease (GvHD)
Description: The cumulative incidence of overall grades II-IV and grades III-IV acute GVHD will be assessed through six months after last dose of FMT or placebo. Acute GVHD will be assessed using the Mount Sinai Acute GVHD International Consortium (MAGIC) criteria.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | FMT Capsules | Placebo Capsules
Number analyzed (Participants) | 3 | 3
Participants | 2 | 0

3. Secondary Outcome: Number of Participants With Non-relapse-mortality
Description: Non-relapse mortality (NRM) is defined as the time from first dose of FMT or placebo to death without relapse or progression or underlying disease.
Time Frame: 6 Months and 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | FMT Capsules | Placebo Capsules
Number analyzed (Participants) | 3 | 3
Participants
  at 6 months | 1 | 0
  at 12 months (cumulative) | 2 | 0

4. Secondary Outcome: Number of Participants With Infection at 100 Days
Time Frame: 100 Days
Measure: Count of Participants; unit: Participants
Arm/Group | FMT Capsules | Placebo Capsules
Number analyzed (Participants) | 3 | 3
Participants | 2 | 0

5. Secondary Outcome: Number of Participants With Progression Free Survival at 12 Months Post-treatment
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Progression-Free Survival (PFS) is defined as the time from first dose of FMT or placebo to the earlier of underlying disease progression or death due to any cause. PFS was assessed at 12 months for all participants.
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | FMT Capsules | Placebo Capsules
Number analyzed (Participants) | 3 | 3
Participants | 1 | 1

6. Secondary Outcome: Overall Survival
Description: Overall survival is measured as the amount of time from the first dose of Fecal Microbiota Transplantation (FMT) or placebo, that participants in this study are still alive. Overall survival is reported as number of participants alive at 12 months.
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | FMT Capsules | Placebo Capsules
Number analyzed (Participants) | 3 | 3
Participants | 1 | 2

7. Secondary Outcome: Graft Versus Host Disease(GVHD)/ Relapse Free Survival (GRFS)
Description: GVHD-Free/Relapse-Free Survival (GRFS) is measured as the amount of time from the first dose of Fecal Microbiota Transplantation (FMT) or placebo, that participants in this study are not diagnosed with GVHD, disease progression, or relapse. GRFS is reported as number of patients without GVHD, disease progression, or relapse at 12 months.
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | FMT Capsules | Placebo Capsules
Number analyzed (Participants) | 3 | 3
Participants | 0 | 2

ADVERSE EVENTS:
Time Frame: Adverse event data collection time frame was approximately 13 months, starting 1 week after allogeneic hematopoietic cell transplantation (HCT) until 12 months after the second fecal microbiota transplantation (FMT) or placebo administration.
Arm/Group | FMT Capsules | Placebo Capsules
All-Cause Mortality (participants affected / at risk) | 2/3 | 1/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FMT Capsules (N=3) | Placebo Capsules (N=3)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FMT Capsules (N=3) | Placebo Capsules (N=3)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Neutrophil count decreased (Investigations) | 2 | 1
Platelet count decreased (Investigations) | 2 | 3
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-11): https://cdn.clinicaltrials.gov/large-docs/92/NCT03720392/Prot_SAP_000.pdf